CLINICAL TRIAL: NCT02915653
Title: Adult Primary and Preventive Practice (APPP) Study
Acronym: APPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Collaborators: Applied Proteomics Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Pro000018813
Record Dates: First submitted 2016-09-22; First posted 2016-09-27 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Preventive Care

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Control: not receiving any intervention
- Intervention 1 (Experimental): Receiving educational materials on a new diagnostic service
  Interventions: Other: Educational materials on a new diagnostic service
- Intervention 2 (Experimental): Receiving educational materials on a new diagnostic service
  Interventions: Other: Educational materials on a new diagnostic service

INTERVENTIONS:
Other: Educational materials on a new diagnostic service — Educational materials on a new diagnostic service
  Arms: Intervention 1; Intervention 2

SUMMARY:
The study is a pre-post two round, randomized controlled study design of PCPs randomly assigned to a control or 1 of 2 intervention arms.

ELIGIBILITY:
Inclusion Criteria:

* 1. Provide consent to participate in the study 2. Board-certified physician currently practicing in the following areas: 3. Internal medicine 4. Family medicine 5. Have practiced as a board-certified physician in internal or family medicine for greater than 2 but less than 30 years. 6. English-speaking 7. Community / non-academic based practice setting 8. ≥ 40 patients under care weekly 9. Access to the internet

Exclusion Criteria:

* 1. Not board certified in their respective area of care 2. Academic-based practice 3. Have practiced as a board-certified physician for less than 2 or greater than 30 years 4. Follow <40 patients weekly 5. Non-English speaking 6. Unable to access the internet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Quality of Care | 8 weeks
  Difference in difference of combined diagnostic and treatment CPV domain scores, including colonoscopy referral rates, in post-intervention versus baseline comparing intervention and control groups among the three patient types.

SECONDARY OUTCOMES:
Intervention Impact on Care | 8 weeks
  Difference in difference between the control and intervention groups in the overall quality of care for CRC screening and for adult primary prevention care measured by the combined and individual item CPV scores for the three patient types.
Healthcare Utilization | 8 weeks
  Difference in health care utilization and/or costs in patients tested with SimpliPro Colon™ versus the control group.
Diagnostic Method Comparison | 8 weeks
  Difference in recommendation of CRC evaluation with colonoscopy and/or flexible sigmoidoscopy, double barium enema, or CT colonography, including risk-level and urgency pre- and post-intervention, between intervention and control groups

CONTACTS AND LOCATIONS:
Overall Officials: John Peabody, MD, PhD, Principal Investigator — QURE Healthcare
Locations (1):
- QURE Healthcare, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No